CLINICAL TRIAL: NCT06635512
Title: The Effect of Stress Ball Application After Transurethral Resection of the Prostate on Patients' Recovery Quality and Hospital Discharge Time: A Randomized Controlled Study
Brief Title: The Effect of Stress Ball on Recovery Quality and Hospital Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seval Ulubay (Other)
Responsible Party: Sponsor-Investigator, Seval Ulubay, PhD, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUR
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Stress
Keywords: stress ball; Recovery quality; hospital discharge; the effect of stress ball

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Ball Impact on Post-Transurethral Resection Recovery. (Experimental): Participants will use stress balls regularly, and outcomes such as physical strength, pain levels, and psychological well-being will be assessed to evaluate the intervention's impact.
  Interventions: Other: The Effect of Stress Ball Application After Transurethral Resection of the Prostate on Patients' Recovery Quality and Hospital Discharge Time
- The effect of the stress ball on patients' discharge time. (Experimental): This arm of the study examines how the use of stress balls during recovery affects the length of hospital stay and discharge time for patients
  Interventions: Other: The Effect of Stress Ball Application After Transurethral Resection of the Prostate on Patients' Recovery Quality and Hospital Discharge Time

INTERVENTIONS:
Other: The Effect of Stress Ball Application After Transurethral Resection of the Prostate on Patients' Recovery Quality and Hospital Discharge Time — The effect of the stress ball applied after surgery on patients' recovery quality will be evaluated.
  Other Names: To examine the effects of the stress ball after surgery.

SUMMARY:
This study aims to investigate the effect of stress ball application after transurethral resection of the prostate on patients' recovery quality and hospital discharge time.

DETAILED DESCRIPTION:
The stress ball, one of the distraction methods, is an effective technique for ensuring cognitive focus. It has been observed that the stress ball method is used to reduce patients' anxiety and pain. Squeezing a stress ball during a surgical procedure allows patients to have direct control over the object, enhancing their feelings of empowerment. In this way, it positively impacts anxiety and patient satisfaction without interfering with the surgical process. In the study by Yanes et al., the effects of the stress ball and hand-holding on pain, anxiety, and satisfaction were evaluated during skin cancer surgery performed under local anesthesia. Although anxiety was observed to decrease in all groups, no significant difference was found between the groups regarding pain and anxiety. It was noted that nearly all participants were very satisfied. The use of the stress ball appears to help reduce anxiety in anxious patients prior to the procedure. In a study conducted by Kasar et al. on hemodialysis patients, the effects of stress ball usage on stress, vital signs, and comfort levels were investigated. While the use of the stress ball did not affect vital signs and comfort, it demonstrated a positive impact on stress. In a study investigating the effects of distraction methods used during cystoscopy on pain, anxiety, and satisfaction, it was found that anxiety levels post-procedure were lower in the intervention groups (music, video, and stress ball) compared to the control group, while satisfaction levels were higher . Another randomized controlled study evaluated the effectiveness of three different non-pharmacological methods (coughing technique, spirometer blowing, and squeezing a stress ball) in reducing pain during intravenous catheterization. It was reported that the average pain levels in the coughing, spirometer, and stress ball groups were lower compared to the control group . In a study examining the effectiveness of distraction methods for pain and anxiety management during invasive venous surgical procedures, it was indicated that pain and anxiety levels were significantly lower in the interaction with nurses and stress ball group . In a study on managing dental anxiety with the application of a stress ball, no significant difference was found between the anxiety scores of patients who used the stress ball and those who did not. Similarly, in another study investigating the effects of distraction methods during lithotripsy, no significant difference was observed in pain and anxiety scores between the control and intervention groups (music and stress ball) .

ELIGIBILITY:
Inclusion Criteria:

Will be applied to patients who are over 18 years old. Have no hearing or vision problems. Can read and write, and can communicate effectively.

Exclusion Criteria:

Patients under 18 years of age. Patients with communication problems.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
The effect of the method used on post-surgery recovery quality | 10 weeks
  The primary outcome measure for this study will be the overall quality of post-surgery recovery, assessed through standardized questionnaires evaluating functional mobility, and patient satisfaction

SECONDARY OUTCOMES:
The effect of the stress ball applied after surgery on patients' discharge time will be evaluated. | 10 weeks
  The primary outcome measure will be the difference in discharge times between patients who used stress balls post-surgery and those who did not.

CONTACTS AND LOCATIONS:
Overall Officials: Seval ULUBAY, PHD, Principal Investigator — Samsun Gazi State Hospital
Locations (1):
- Seval Ulubay, Samsun, Atakum/Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
This IPD Sharing Plan investigates the impact of stress ball application on recovery quality and hospital discharge time after transurethral resection of the prostate (TURP). Conducted by the Department of Urology at a University Hospital, it involves researchers, data analysts, and patients in intervention and control groups. The plan outlines clear roles, promotes collaboration, and ensures equitable sharing of findings. Weekly meetings and regular reports will facilitate communication, while performance metrics will assess recovery outcomes. Ongoing training will enhance ethical standards and data collection, aiming to optimize patient recovery through transparent stakeholder collaboration.
Supporting Information: Study Protocol
Time Frame: 24 WEEKS
Access Criteria: The access criteria for this study on stress ball application post-TURP establish clear inclusion and exclusion guidelines. Eligible participants are adult males aged 50 and older with benign prostatic hyperplasia (BPH) who can provide informed consent. Exclusion criteria include prior prostate surgeries, severe comorbidities, cognitive impairments, and allergies to stress ball materials. Data access is limited to the research team and the Clinical Ethics Committee to ensure ethical oversight and confidentiality through data anonymization. Participants may withdraw at any time without penalty. Collected data will be securely stored, with compliance monitored to uphold ethical standards and protect patient confidentiality during the evaluation of the stress ball application's effectiveness.